CLINICAL TRIAL: NCT00717366
Title: An Open-Label Multi-center, Multiple Dose Study to Determine the Optimum Starting Dose of Intravenous MIRCERA for Maintenance Treatment of Anemia in Pediatric Participants With Chronic Kidney Disease on Hemodialysis
Brief Title: Study to Determine Optimum Intravenous Starting Dose of MIRCERA for Treatment of Pediatric Participants With Anemia and Chronic Kidney Disease on Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH19707; 2007-007758-70 (EudraCT Number)
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Renal Anemia
MeSH Terms: interventions — continuous erythropoietin receptor activator

ARMS (2):
- MIRCERA Group 1: Intermediate-Conversion-Factor Group (Experimental): Participants will receive methoxy polyethylene glycol-epoetin beta (MIRCERA) IV injection at a starting dose based on an intermediate conversion factor from their previous Erythropoiesis-stimulating Agent (ESA) dose (4 * previous weekly epoetin dose [international units {IU}]/250 or 4 * previous weekly darbepoetin alfa dose [micrograms {mcg}]/1.1) once every 4 weeks for 20 weeks. Participants who will complete the 20 weeks of treatment with hemoglobin (Hb) level within ± 1 grams per deciliter (g/dL) of their baseline Hb level and within the target range of 10-12 g/dL will enter an optional 52-weeks safety extension period. During this period, the participants will continue to receive MIRCERA IV injection once every 4 weeks.
  Interventions: Drug: Methoxy Polyethylene Glycol-Epoetin Beta
- MIRCERA Group 2: High-Conversion-Factor Group (Experimental): Participants will receive MIRCERA IV injection based on a high conversion factor from their previous ESA dose (4 * previous weekly epoetin dose [IU]/125 or 4 * previous weekly darbepoetin alfa dose [mcg]/0.55) once every 4 weeks for 20 weeks. Participants who will complete the 20 weeks of treatment with Hb within ± 1 g/dL of their baseline Hb and within the target range of 10-12 g/dL will enter an optional 52-weeks safety extension period. During this period, the participants will continue to receive MIRCERA IV injection once every 4 weeks.
  Interventions: Drug: Methoxy Polyethylene Glycol-Epoetin Beta

INTERVENTIONS:
Drug: Methoxy Polyethylene Glycol-Epoetin Beta — Will be administered IV, every 4 weeks.
  Other Names: MIRCERA; RO0503821

SUMMARY:
This sequential study will assess the efficacy and safety of multiple doses of intravenous (IV) methoxy polyethylene glycol-epoetin beta (MIRCERA), and will determine the optimum starting dose for maintenance treatment of anemia in children with chronic kidney disease on hemodialysis. Pediatric participants will remain on epoetin alfa, epoetin beta or darbepoetin alfa during the screening period, after which they will receive IV MIRCERA monthly, at a starting dose related to the previous weekly epoetin or darbepoetin alfa dose. Depending on the response achieved, another group may be selected to receive a higher or a lower dose.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-17 years (in Russia only: 12-17 years) with clinically stable chronic renal anemia
* Hemodialysis for greater than or equal to (>=) 8 weeks
* Intravenous stable maintenance treatment with epoetin alfa, epoetin beta, or darbepoetin alfa for >= 8 weeks before screening and with no weekly dose change >= 25 percent (%) (increase or decrease) during the 2 weeks of screening

Exclusion Criteria:

* Overt gastrointestinal bleeding within 8 weeks before screening or during the screening period
* Red blood cell (RBC) transfusions within 8 weeks before screening or during the screening period
* Active malignant disease
* Pure red cell aplasia (PRCA) or history of PRCA
* Pregnant or lactating females
* Sexually active participants: not willing to use reliable contraception during treatment and for 90 days following the end of treatment

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- Royal Children'S Hospital; Department of Nephrology, Parkville, Victoria, Australia
- Belgium (2):
  - Hôpital Enfants Reine Fabiola, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- France (7):
  - Hopital Femme Mere Enfant; Ped Nephrologie Rhumatologie, Bron
  - Hopital Jeanne De Flandre; Cons Pediatrie, Lille
  - Hopital Timone Enfants; Nephrologie Hemodialyse, Marseille
  - Hopital Arnaud De Villeneuve; Pediatrie I, Montpellier
  - Hôpital Robert Debré; Nephrologie pediatrique, Paris
  - Hopital Armand Trousseau; Pediatrie Nephrologie, Paris
  - Höpital Hautepierre; Pediatrie 1, Strasbourg
- Germany (5):
  - Klinik der Uni zu Köln; Kinderklinik, Cologne
  - KfH Nierenzentrum für Kinder und Jugendliche, Hamburg
  - KfH-Nierenzentrum fur Kinder und Jugendliche, Heidelberg
  - Kinderklinik Memmingen; Kinderdialysezentrum, Memmingen
  - KfH-Nierenzentrum für Kinder und Jugendliche, Münster
- Semmelweis University; 1st Department of Pediatrics, Pediatric Nephrology Center, Budapest, Hungary
- Italy (4):
  - Ospedale Pediatrico Bambino Gesu; U.O. Di Nefrologia E Dialisi, Rome, Lazio
  - IRCCS G. Gaslini; U.O. Nefrologia, Dialisi e Trapianto, Genoa, Liguria
  - Ospedale Infantile Regina Margherita; U.O. Autonoma di Nefrologia, Dialisi e Trapianto, Turin, Piedmont
  - A.O. Di Padova; Dipartimento Di Pediatria U.O. Di Nefrologia Pediatrica, Dialisi e Trapianto, Padua, Veneto
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne; Klinika Chorob Nerek i Nadciśnienia Dzieci i Mlodziezy, Gdansk
  - Instytut "Centrum Zdrowia Matki Polki; Klinika Nefrologii i Dializoterapii, Lodz
  - Dzieciecy Szpital Kliniczny; Klinika Nefrologii Dzieciecej, Lublin
  - SPSZOZ Zdroje Oddzial Pediatrii; Nefrologii i Toksykologii ze Stacja Dializ, Szczecin
  - Wojewodzki Szpital Dzieciecy; Osrodek Chorob Nerek i Dializoterapii, Torun
  - Instytut Pomnik-Centrum Zdrowia Dziecka, Klinika Nefrologii, Transp. Nerek i Nadcisnienia Tetniczego, Warsaw
  - Akademia Medyczna im. Piastow Slaskich; Katedra i Klinika Nefrologii Pediatrycznej, Wroclaw
- Romania (2):
  - Fundeni Clinical Institute, Bucharest
  - St. Maria Emergency Clinical Hospital for Children, Iași
- Russia (2):
  - DGCB St. Vladimir; Pediatric nephrologist, Moscow
  - SBIH Children City Hospital #1; Dialysis department, Saint Petersburg
- Spain (4):
  - Hospital Universitari Vall d'Hebron; Servicio de Nefrologia, Barcelona
  - Hospital Universitario La Paz: Nefrologia Pediatrica, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Nefrologia Pediatrica, Seville
  - Hospital Universitario la Fe; Servicio de Nefrologia Pediatrica, Valencia
- Thailand (2):
  - Chulalongkorn university Faculty of Medicine;Department of Pediatrics, Bangkok
  - Siriraj Hospital, Faculty of Medicine; Department of Pediatrics, Bangkok
- Ukraine (2):
  - Kiev city childrens nephrological center of hospital #1; Nephrology and RRT, Kiev
  - Public Institution Zaporizhzhia City Multispecialty Children's Hospital #5; Allergologic, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 112 participants were screened at 28 sites in 10 countries, of which 64 participants were enrolled (16 initially in MIRCERA Group 1 and then 48 in MIRCERA Group 2, following a preliminary analysis of MIRCERA Group 1).
Groups:
- MIRCERA Group 1: Intermediate-Conversion-Factor Group: Participants received methoxy polyethylene glycol-epoetin beta (MIRCERA) intravenous (IV) injection at a starting dose based on an intermediate conversion factor from their previous Erythropoiesis-Stimulating Agent (ESA) dose (4 * previous weekly epoetin dose [international units {IU}]/250 or 4 * previous weekly darbepoetin alfa dose [micrograms {mcg}]/1.1) once every 4 weeks for 20 weeks. Participants who completed the 20 weeks of treatment and had hemoglobin (Hb) level within ± 1 grams per deciliter (g/dL) of their baseline Hb level and within the target range of 10-12 g/dL, entered an optional 52-weeks safety extension period. During this period, the participants continued to receive MIRCERA IV injection once every 4 weeks.
- MIRCERA Group 2: High-Conversion-Factor Group: Participants received MIRCERA IV injection based on a high conversion factor from their previous ESA dose (4 * previous weekly epoetin dose [IU]/125 or 4 * previous weekly darbepoetin alfa dose [mcg]/0.55) once every 4 weeks for 20 weeks. Participants who completed the 20 weeks of treatment and had Hb level within ± 1 g/dL of their baseline Hb level and within the target range of 10-12 g/dL, entered an optional 52-weeks safety extension period. During this period, the participants continued to receive MIRCERA IV injection once every 4 weeks.
Period: Core Study Period (20 Weeks)
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Started | 16 | 48
Completed | 12 | 35
Not Completed | 4 | 13
Not completed — Renal transplant | 4 | 9
Not completed — Admin/Other than specified | 0 | 2
Not completed — Death | 0 | 1
Not completed — Refused treatment/Did not cooperate | 0 | 1
Period: Extension Period (52 Weeks)
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Started | 9 | 28
Received Visit/Week 21 Dose | 8 | 28
Completed | 5 | 12
Not Completed | 4 | 16
Not completed — Renal transplant | 3 | 13
Not completed — Admin/Other than specified | 0 | 2
Not completed — Withdrew consent | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all enrolled participants.
Groups:
- MIRCERA Group 1: Intermediate-Conversion-Factor Group: Participants received MIRCERA IV injection at a starting dose based on an intermediate conversion factor from their previous ESA dose (4 * previous weekly epoetin dose [IU]/250 or 4 * previous weekly darbepoetin alfa dose [mcg]/1.1) once every 4 weeks for 20 weeks. Participants who completed the 20 weeks of treatment and had Hb level within ± 1 g/dL of their baseline Hb level and within the target range of 10-12 g/dL, entered an optional 52-weeks safety extension period. During this period, the participants continued to receive MIRCERA IV injection once every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group | Total
Number analyzed (Participants) | 16 | 48 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (3.24) | 13.0 (3.06) | 12.6 (3.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 25 | 30
  Male | 11 | 23 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Hb Concentration Between Baseline and Evaluation Period
Description: A time adjusted average baseline Hb concentration for each individual was calculated using an area under the curve (AUC) approach from all available Hb measurements taken during the baseline period (Day -20 to Day 1). The average evaluation period Hb concentration for each individual was calculated using the same method, from all their available measurements taken during the evaluation period (Week 17 to Week 21). The change in Hb concentration between the baseline and evaluation periods was calculated by subtracting the baseline Hb concentration from the evaluation period Hb concentration.
Time Frame: Baseline (Day -20 to Day 1), Evaluation Period (Week 17 to Week 21)
Population: ITT population. Hb values within 21 days after blood transfusion(s) were excluded from analysis.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Number analyzed (Participants) | 16 | 48
g/dL
  Baseline (n=16,48) | 11.26 (0.496) | 11.08 (0.493)
  Change at Evaluation Period (n=12,36) | -0.78 (1.237) | -0.15 (1.014)

2. Secondary Outcome: Number of Participants With an Average Hb Concentration During the Evaluation Period Within ±1 g/dL of Their Baseline Hb
Description: Baseline Hb value was defined as the average Hb concentration from all available Hb measurements taken during the baseline period (Day -20 to Day 1). The evaluation period Hb concentration was defined as the average Hb concentration from all available Hb measurements taken during the evaluation period (Week 17 to Week 21).
Time Frame: Evaluation Period (Week 17 to Week 21)
Population: ITT population. Hb values within 21 days after blood transfusion(s) were excluded from analysis. Number of participants analyzed = participants with Hb concentration assessment at specified time-points.
Measure: Number; unit: participants
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Number analyzed (Participants) | 12 | 36
participants | 7 | 27

3. Secondary Outcome: Number of Participants With an Average Hb Concentration During the Evaluation Period Above, Within or Below the Range of 10-12 g/dL
Description: The evaluation period Hb concentration was defined as the average Hb concentration from all available Hb measurements taken during the evaluation period (Week 17 to Week 21).
Time Frame: Evaluation Period (Week 17 to Week 21)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Number analyzed (Participants) | 12 | 36
participants
  Above 12 g/dL | 0 | 3
  Within 10-12 g/dL | 9 | 29
  Below 10 g/dL | 3 | 4

4. Secondary Outcome: Number of Participants With Blood Transfusions
Time Frame: Baseline to Week 20
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Number analyzed (Participants) | 16 | 48
participants | 1 | 2

5. Secondary Outcome: Change in Average Reticulocyte Count Between the Baseline and Evaluation Period
Description: A time adjusted average baseline reticulocyte count for each individual was calculated using an AUC approach from all available reticulocyte counts taken during the baseline period (Day -20 to Day 1). The average evaluation period reticulocyte count for each individual was calculated using the same method, from all their available measurements taken during the evaluation period (Weeks 17 to 21). The change in reticulocyte count between the baseline and evaluation periods was calculated by subtracting the baseline reticulocyte count from the evaluation period reticulocyte count. Relative reticulocytes were recorded conversion to absolute values was performed.
Time Frame: Baseline (Day -20 to Day 1), Evaluation Period (Week 17 to Week 21)
Population: ITT population. Reticulocyte values within 21 days after blood transfusion(s) were excluded from analysis. Here, number of participants analyzed = participants evaluable for this outcome measure and 'n' signifies number of participants evaluable at specified time-points.
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Number analyzed (Participants) | 15 | 48
10^3 cells/microliter
  Baseline (n=15,48) | 46.08 (26.472) | 43.70 (25.984)
  Change at Evaluation Period (n=11,36) | 23.38 (29.279) | 24.80 (32.428)

6. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MIRCERA
Description: Cmax was defined as the highest serum concentration observed from all sample collection timepoints (as provided in timeframe) and was averaged out among participants and reported.
Time Frame: Pre-dose (with 1 hour before drug administration) and 2, 48 hours post dose on Week 9, at Weeks 10, 11, and 12, pre-dose (with 1 hour before drug administration) on Week 13
Population: Pharmacokinetic (PK) evaluable population included all enrolled participants who received at least one dose of study drug and had evaluable PK assessment. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Number analyzed (Participants) | 12 | 34
picograms per milliliter (pg/mL) | 37700 (74.5) | 66100 (149.5)

7. Secondary Outcome: Area Under the Serum Concentration-Time Curve From 0 to 672 Hours (AUC0-672h) of MIRCERA
Description: Area under the serum concentration versus time curve over 672 hours. AUC0-672h represents area under the serum concentration versus time curve from time zero to end of dosing interval (AUC0-tau).
Time Frame: as for outcome 6
Population: PK evaluable population. Number of participants analyzed = participants with AUC0-672h assessment at specified time-points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms*hour/milliliter (pg*h/mL)
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Number analyzed (Participants) | 11 | 32
picograms*hour/milliliter (pg*h/mL) | 3630000 (91.8) | 7170000 (140.0)

8. Secondary Outcome: Time to Reach Cmax (Tmax) of MIRCERA
Description: Tmax was defined as the time (in hours) to achieve Cmax (Cmax was defined as the highest serum concentration observed over all sample collection timepoints [as provided in timeframe]). The median time, among all participants, was reported.
Time Frame: as for outcome 6
Population: PK evaluable population.
Measure: Median (Full Range); unit: hours
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Number analyzed (Participants) | 12 | 34
hours | 2.00 [1.98 to 2.17] | 2.00 [1.83 to 164]

9. Secondary Outcome: Apparent Terminal Phase Half-Life (t1/2) of MIRCERA
Description: t1/2 was defined as the time (in hours) measured (from all sample collection timepoints [as provided in timeframe]) for the serum concentration to decrease by one half. The t1/2 was calculated as natural logarithm of 2 divided by λz; where λz = terminal elimination rate constant.
Time Frame: as for outcome 6
Population: PK evaluable population. Number of participants analyzed = participants evaluable for t1/2 assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Number analyzed (Participants) | 11 | 32
hours | 147 (30.1) | 121 (43.5)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 73
Description: Safety population included all participants who received at least one dose of study drug and had a safety follow-up visit.
Arm/Group | MIRCERA Group 1: Intermediate-Conversion-Factor Group | MIRCERA Group 2: High-Conversion-Factor Group
Serious Adverse Events (participants affected / at risk) | 4/16 | 17/48
Other Adverse Events (participants affected / at risk) | 11/16 | 28/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MIRCERA Group 1: Intermediate-Conversion-Factor Group (N=16) | MIRCERA Group 2: High-Conversion-Factor Group (N=48)
Device related infection (Infections and infestations) | 0 | 3
Bronchitis (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 2
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Thrombosis in device (General disorders) | 0 | 3
Device dislocation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intracranial haematoma (Nervous system disorders) | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MIRCERA Group 1: Intermediate-Conversion-Factor Group (N=16) | MIRCERA Group 2: High-Conversion-Factor Group (N=48)
Nasopharyngitis (Infections and infestations) | 0 | 14
Bronchitis (Infections and infestations) | 1 | 3
Pharyngitis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 1 | 2
Catheter site infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
H1N1 influenza (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 13
Paraesthesia (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 3
Malaise (General disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.